CLINICAL TRIAL: NCT06413121
Title: An Observer-blind, Randomized, Active-controlled, Multi-centric Phase III Study to Assess Immunogenicity and Safety of Hexavalent (DTwP-Hepatitis B-IPV-Hib) Vaccine Containing Reduced Dose IPV in Comparison With HEXASIIL®
Brief Title: Clinical Study to Assess the Immunogenicity and Safety of Hexavalent Vaccine Containing Reduced Dose IPV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SII-wHEXA/IN-03
Record Dates: First submitted 2024-05-03; First posted 2024-05-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diptheria Immunization; Tetanus Immunization; Pertussis Immunization; Hepatitis B Immunization; Haemophilus Influenzae Type B Immunization; Polio Immunization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Reduced Dose IPV (Experimental): Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Reduced Dose IPV for active immunization of infants, as a 3 dose regimen (6, 10 & 14 weeks) for primary vaccination and booster dose at the age of 12-24 months.
  Interventions: Biological: Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Reduced Dose IPV
- Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Full Dose IPV (Active Comparator): Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Full Dose IPV for active immunization of infants, as a 3 dose regimen (6, 10 & 14 weeks) for primary vaccination and booster dose at the age of 12-24 months.
  Interventions: Biological: Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Full Dose IPV

INTERVENTIONS:
Biological: Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Reduced Dose IPV — Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Reduced Dose IPV for active immunization of infants as 3 dose regimen (6, 10 & 14 weeks) for primary vaccination and booster dose at the age of 12-24 months.
  Arms: Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Reduced Dose IPV
Biological: Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Full Dose IPV — Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Full Dose IPV for active immunization of infants as 3 dose regimen (6, 10 & 14 weeks) for primary vaccination and booster dose at the age of 12-24 months.
  Arms: Hexavalent (DTwP-HepB-IPV-Hib) Vaccine Containing Full Dose IPV

SUMMARY:
In 2012, the World Health Assembly (WHA) endorsed the proposed Polio Endgame Strategy, which includes withdrawal of the Sabin-virus type 2 antigen-responsible for an estimated 95% of vaccine derived cases of polio by replacing the trivalent Oral Polio Vaccine (OPV) in the routine immunization schedule with a bivalent OPV that lacks the type 2 Sabin virus. Since the WHA resolution, all countries that were solely using OPV have either introduced Inactivated Polio Vaccine (IPV) into their routine immunization schedule or decided to introduce IPV but have been unable to secure supply. The global demand for IPV has therefore substantially increased in just a few years. Many initiatives are ongoing to meet the increasing demand for IPV. One potential approach is the reduction of the amount of antigen per vaccine dose. Therefore, to enhance the affordability, effectiveness and accessibility of IPV.

SIIPL has manufactured hexavalent combination vaccine containing diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b and a reduced dose of three IPV antigens.

Based on available published data, reduction of the antigen content of each of the three poliovirus types in IPV is feasible, without substantially compromising the immunogenicity of the vaccine. Advantages of a reduction in antigen content are two-fold: increased availability of IPV and reduced cost, both of major importance for the global eradication programme.

DETAILED DESCRIPTION:
This is an observer-blind, randomized, active-controlled, multi-centric study in healthy infants and toddlers to assess the immunogenicity and safety of SIIPL reduced IPV hexavalent vaccine in comparison with the licensed SIIPL HEXASIIL® vaccine.

One thousand five hundred and fifty-seven infants aged 6-8 weeks (42 to 56 days, both days inclusive) will be randomized in a 2:1 ratio (1038 infants in SIIPL reduced IPV hexavalent group and 519 in SIIPL HEXASIIL® group), to receive a 3-dose primary vaccination series followed by their booster doses, respectively. The safety and immunogenicity data collected up to 28 days following third vaccination i.e., Visit 7, shall be submitted to the regulatory authority. All subjects will be followed up further for booster dose. After Visit 7 (i.e., 28 days following completion of primary vaccination series) subjects will be followed up for safety every 3 months starting from the age of 6 months (i.e., at 6, 9, 12, 15, 18, and 21 months of age) until they receive the booster dose anytime between 12-24 months. There will be post booster follow up visit (EOS visit) 28 days after the booster immunization i.e., Visit 10 to assess the safety and post booster immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants aged 6-8 weeks at the time of first vaccination.
* Infants with good health, as determined by the medical history, physical examination and clinical judgment of the Investigator.
* Informed consent form signed by at least one parent.
* Infants born at full term pregnancy (≥ 37 weeks).
* Infants with weight-for-length z-score ≥ -2 standard deviation (SD) at the time of enrolment.
* Willingness of subjects' parent to comply with the requirements of the protocol.

Exclusion Criteria:

* History of diphtheria/ tetanus/ pertussis/ hepatitis B/ Haemophilus Influenzae type b/ poliomyelitis infection(s).
* Presence of fever ≥ 38°C/ 100.4°F.
* Acute illness of moderate to severe intensity according to the clinical judgment of the investigator .
* Receipt of antibiotics in the past 3 days
* Previous vaccination or planned receipt of any vaccine against diphtheria, tetanus, pertussis, hepatitis B (except birth dose), poliomyelitis (except OPV birth dose) or Haemophilus Influenzae type b infection apart from trial vaccines during the study period.
* Administration of any vaccine (except OPV during government immunization campaign) in the 4 weeks preceding the first trial vaccination.
* History of major congenital defects or illness that require medical therapy, as determined by medical history or clinical assessment.
* History of any clinically significant chronic disease that in the opinion of the Investigator, might interfere with the evaluation of the study objectives.
* History of anaphylaxis, or any serious vaccine reaction, or hypersensitivity/allergy to any vaccine or components of study vaccine.
* Infants with known or suspected impairment of the immune function, or those receiving immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy or received immunosuppressive therapy prior to study entry
* Presence of evolving or changing neurological disorder or infant with a history of seizures and/or encephalopathy.
* Known thrombocytopenia or a bleeding disorder.
* Known personal or maternal history of HIV, Hepatitis B or Hepatitis C seropositivity.
* Planned surgery during the study.
* Receipt of blood or blood-derived products or immunoglobulins or planned administration during the trial which might interfere with the assessment of the immune response.
* Participation in another clinical trial 4 weeks preceding the trial enrolment or planned participation during the present trial period in another clinical trial.
* Infants whose families are planning to leave the area of the study site before the end of the study period.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1557 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of SIIPL reduced IPV hexavalent vaccine in comparison with SIIPL HEXASIIL® vaccine. | 28 days post completion of 3-dose primary vaccination series in infants.
  Percentage of infants achieving seroprotection for diphtheria, tetanus, hepatitis B, Haemophilus influenzae type b, poliovirus types 1, 2 & 3, seroresponse for anti-B. pertussis and seroconversion for anti-pertussis toxin, 28 days post completion of a 3-dose primary vaccination series.

SECONDARY OUTCOMES:
Assessment of occurrence, severity, and relationship of adverse events (AEs) | Local and systemic solicited AEs occurring up to 7 days following each vaccination, unsolicited AEs and SAEs till 28 days post completion of a 3-dose primary vaccination series.
  local and systemic solicited AEs, unsolicited AEs and serious adverse events (SAEs)
Assessment of immunogenicity of SIIPL reduced IPV hexavalent vaccine with the comparator vaccine, SIIPL HEXASIIL® and to assess lot-to-lot consistency among 3 lots of SIIPL reduced IPV Hexavalent vaccine | 28 days post completion of the 3-dose primary vaccination series in infants.
  Geometric mean concentrations/ Geometric mean titres (GMCs/GMTs) for anti diphtheria, anti-tetanus, anti-B. pertussis, anti-pertussis toxin, anti-HBsAg, anti- polyribosylribitol phosphate (PRP) and anti-polio types 1, 2 & 3 antibodies, 28 days post completion of the 3 dose primary vaccination series in infants.

OTHER OUTCOMES:
Pre- and post-booster safety of SIIPL reduced IPV hexavalent vaccine and comparator vaccine, SIIPL HEXASIIL® in toddlers. | Safety assessment from 28 days post completion of the 3-dose primary schedule till 28 days post booster.
  Local and systemic solicited AEs occurring up to 7 days and unsolicited AEs and SAEs till 28 days post completion of booster vaccination.
Pre- and post-booster immunogenicity of SIIPL reduced IPV hexavalent vaccine and comparator vaccine, SIIPL HEXASIIL® in toddlers. | Immunogenicity at prebooster and 28 days post booster dose between 12-24 months of age.
  GMTs/ GMCs and Percentage of toddlers achieving seroprotection/seroconversion for diphtheria, tetanus, hepatitis B, Haemophilus influenzae type b, poliovirus types 1, 2 & 3 and pertussis, prior to booster dose and 28 days after a booster dose.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kawade, Principal Investigator — KEM Hospital Research Centre, Pune, India; Sonali Palkar, Principal Investigator — Bharati Vidyapeeth Medical College Hospital and Research Centre, Pune, India; M D Ravi, Principal Investigator — JSS Hospitla, Mysore, India; Veena Kamat, Principal Investigator — Manipal Academy of Higher Education, Kasturba Medical College, Udipi and Karkala,India; P Umapathy, Principal Investigator — Sri Ramchndra Institute of Higher Education and Research, Chennai, India; Kheya Ghosh, Principal Investigator — Institute of Child Health, Kolkata, India; Madhu Gupta, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh, India; Afreen khan, Principal Investigator — Hamdard Institute of Medical Sciences and Research (HIMSR), New Delhi, India; Deepali Ambike, Principal Investigator — Yashwantrao Chavan Memorial Hospital, Pimpri, Pune, India; K Zaman, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh
Locations (9):
- International Centre for Diarrhoeal Disease Research, Bangladesh (ICDDR,B), Dhaka, Bangladesh
- India (8):
  - Manipal Academy of Higher Education, Manipal, Mangalore, Karnataka
  - JSS Medical College and Hospital, Mysore, Karnataka
  - Bharati Vidyapeeth Medical College and Hospital, Pune, Pune, Maharashtra
  - KEM Hospital and Research Centre, Vadu, Pune, Maharashtra
  - Hamdard Institute of Medical Sciences and Research (HIMSR) with Centre for health research & Development, Society for applied studies, Hakeem Abdul Hameed Centenary Hospital (HAHCH), New Delhi, National Capital Territory of Delhi
  - Sri Ramachandra Medical Centre, Chennai, Chennai, Tamil Nadu
  - Institute of Child Health, Kolkata, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh

IPD SHARING:
Plan to Share IPD: Yes
Summary results for primary and secondary objectives
Supporting Information: Study Protocol
Time Frame: 6 months after the study completion
Access Criteria: Researchers who provide a methodologically sound proposal may be provided the access afterSponsor permission and if signed data-access agreements are in place.